CLINICAL TRIAL: NCT01027728
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase I/II Study to Evaluate the Safety and Efficacy of CCX354-C in Subjects With Rheumatoid Arthritis
Brief Title: Study to Evaluate Safety and Efficacy of CCX 354-C in Subjects With Rheumatoid Arthritis
Acronym: CARAT-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CL003_354
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CCX354-C (Experimental)
  Interventions: Drug: CCX 354-C

INTERVENTIONS:
Drug: CCX 354-C — * Cohort 1: Eight subjects will be randomized to receive 100 mg CCX354-C or placebo in a ratio of 3:1 (CCX354-C:placebo) once daily for 14 days;
  * Cohort 2: Eight subjects will be randomized to receive 100 mg CCX354-C or placebo in a ratio of 3:1 (CCX354-C:placebo) twice daily for 14 days; and
  * Cohort 3: Eight subjects will be randomized to receive 200 mg CCX354-C or placebo in a ratio of 3:1 (CCX354-C:placebo) once daily for 14 days.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of multiple oral doses of CCX354-C at a number of dose levels in subjects with stable rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled Phase I/II study will consist of two sequential stages, Stage A and B. This protocol describes the objectives, design, and procedures for Stage A of the study. The protocol will be amended in future when sufficient data from Stage A have been collected to initiate Stage B. The protocol amendment will describe the objectives, design, and procedures for Stage B of the study.

Stage A will be a randomized, double-blind, placebo-controlled, multi-dose, sequential dose escalation sub-study in 24 subjects with stable RA. Three sequential dose cohorts of 8 subjects will be included in this stage:

* Cohort 1: 100 mg CCX354-C or placebo
* Cohort 2: 100 mg CCX354-C or placebo
* Cohort 3: 200 mg CCX354-C or placebo

Safety and PK data from each cohort will be reviewed by a data monitoring committee (DMC)before dose escalation to the next dose level. The study will proceed to Stage B only if the safety and tolerability profile of Stage A is deemed acceptable by the DMC.

Study acquired by Amgen and all disclosures were done by previous sponsor ChemoCentryx.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, aged 18-75 years inclusive, with stable RA based on American College of Rheumatology (ACR) criteria (see section 11.3) for at least 3 months (subjects do not need to have active RA for Stage A of the study);
2. Subjects must have been on a stable dose of methotrexate (7.5 to 25 mg/week) taken orally, subcutaneously, or intramuscularly, but not intravenously, for ≥ 8 weeks prior to randomization;
3. If a subject is also taking sulfasalazine or hydroxychloroquine, the subject must have been on a stable dose of these medications for at least 8 weeks prior to randomization;
4. If a subject is on corticosteroid therapy, the dose must not exceed 10 mg prednisone or equivalent and the subject must have been on a stable dose for at least 4 weeks prior to randomization;
5. Willing and able to give written Informed Consent and to comply with the requirements of the study protocol;
6. Negative result of the human immunodeficiency virus (HIV) screen, the hepatitis B screen, and the hepatitis C screen;
7. Judged to be otherwise healthy by the Investigator, based on medical history, physical examination (including electrocardiogram [ECG]), and clinical laboratory assessments;
8. Female subjects of childbearing potential, and male subjects with partners of childbearing potential, may participate if adequate contraception is used during, and for at least the four weeks after, any administration of study medication. Adequate contraception is defined as usage by at least one of the partners of a barrier method of contraception, together with usage by the female partner, commencing at least three months prior to Screening, of a stable regimen of any form of hormonal contraception or an intra-uterine device. Use of abstinence alone is not considered adequate. Use of a barrier method alone is considered adequate only if the male partner was vasectomized at least six months prior to Screening. Use of a double-barrier method of contraception is acceptable.

Exclusion Criteria:

1. Diagnosed with RA prior to 16 years of age;
2. Women who are pregnant, breastfeeding, or have a positive serum pregnancy test at Screening;
3. History within one year prior to randomization of illicit drug use;
4. History of alcohol abuse at any time in the past;
5. Use of infliximab, adalimumab, abatacept, certolizumab, golimumab, or tocilizumab within 8 weeks of randomization;
6. Use of leflunomide within 6 months of randomization;
7. Use of etanercept or anakinra within 4 weeks of randomization;
8. Use of rituximab or ocrelizumab, or cytotoxic agents, such as cyclophosphamide or chlorambucil, within one year of randomization;
9. Currently taking cytochrome P450 inhibitors including protease inhibitors such as ritonavir,indinavir, nelfinavir, or macrolide antibiotics such as erythromycin, telithromycin,clarithromycin, or azole antifungals such as fluconazole, ketoconazole, itraconazole, or cimetidine, nefazodone, bergamottin (constituent of grapefruit juice), quercetin, aprepitant,or verapamil;
10. History or presence of any form of cancer within the 10 years prior to randomization, with the exception of excised basal cell or squamous cell carcinoma of the skin, or cervical carcinoma in situ or breast carcinoma in situ that has been excised or resected completely and is without evidence of local recurrence or metastasis;
11. Evidence of tuberculosis based on chest X rays, tuberculin skin test, QuantiFERON®-TB Gold test, or T-SPOT®.TB test performed during screening;
12. Presence of Felty's syndrome, psoriatic arthritis, or other auto-immune diseases;
13. Major surgery (including joint surgery) within 12 weeks prior to randomization;
14. Subject's hemoglobin is less than 11 g/dL (6.83 mmol/L) at Screening;
15. Subject has any evidence of hepatic disease; AST, ALT, alkaline phosphatase, or bilirubin > 1.5 x the upper limit of normal;
16. Subject has any evidence of renal impairment; serum creatinine > 1.5 x upper limit of normal;
17. The subject had an infection requiring antibiotic treatment within 4 weeks of randomization;
18. History or presence of any medical or psychiatric condition or disease, or laboratory abnormality that, in the opinion of the Investigator, may place the subject at unacceptable risk for study participation and may prevent the subject from completing the study; and
19. Participated in any clinical study of an investigational product within 30 days prior to randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Subject Incidence of Adverse Events | 14 Days

SECONDARY OUTCOMES:
Evaluate possible interaction with methotrexate at a number of dose levels in subjects with stable RA | 14 Days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (5):
- Belgium (2):
  - Brussels
  - Liège
- Romania (3):
  - Bacau
  - Bucharest
  - Galati